CLINICAL TRIAL: NCT06414317
Title: A Comprehensive Education and Navigational Support Program for Advanced Bladder Cancer
Brief Title: An Education and Navigation Support Tool to Improve Participation in Care Coordination Among Patients With Locally Advanced, Metastatic and Unresectable Bladder Cancer and Their Caregivers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: I-3368823; NCI-2024-03446 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I-3368823 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2024-05-06; First posted 2024-05-16 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Locally Advanced Bladder Carcinoma; Metastatic Bladder Carcinoma; Stage III Bladder Cancer AJCC v8; Stage IV Bladder Cancer AJCC v8; Unresectable Bladder Carcinoma
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Nutrition Assessment; Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Supportive Care (ENST) (Experimental): Patients and caregivers receive access to the bladder cancer ENST and patients undergo psychological distress and nutrition screenings and may attend social work, psychology, and/or nutrition consultations as appropriate throughout the study. Patients, caregivers, and providers also attend virtual support group meetings periodically on study.
  Interventions: Procedure: Assessment of Distress; Other: Consultation Visit; Other: Nutritional Assessment; Other: Questionnaire Administration; Other: Supportive Care

INTERVENTIONS:
Procedure: Assessment of Distress — Undergo psychological distress screening
  Other Names: Assessment of Psychological Distress; Evaluation of Patient's Distress
Other: Consultation Visit — Attend consultations
Other: Nutritional Assessment — Undergo malnutrition screening
  Other Names: Dietary Assessment; dietary counseling; nutritional counseling
Other: Questionnaire Administration — Ancillary studies
Other: Supportive Care — Receive access to bladder cancer ENST
  Other Names: Supportive Therapy; Symptom Management; Therapy, Supportive
Other: Supportive Care — Attend virtual support group meetings
  Other Names: Supportive Therapy; Symptom Management; Therapy, Supportive

SUMMARY:
This clinical trial evaluates the impact of an education and navigation support tool (ENST) on patient and caregiver participation in care coordination for bladder cancer that has spread to nearby tissue or lymph nodes (locally advanced), to other places in the body (metastatic) or that cannot be removed by surgery (unresectable). Patients with advanced bladder cancer tend to be older, have multiple medical conditions and often have poor access to health care. An ENST may be an effective method to improve participation in treatment decision-making and care planning among patients with locally advanced, metastatic and unresectable bladder cancer and their caregivers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess project readiness and barriers and requirements to assure success we will evaluate organizational readiness and implementation climate through stakeholder engagement.

II. Development of an ENST to meet the needs of patients and caregivers, the delivery of which is deemed feasible based on such pre-implementation assessment.

III. Implementation and delivery of the proposed ENST. IV. Facilitation of enhanced care coordination for patients with advanced bladder cancer who often have complex medical needs, using measures elaborated in the design and methods section.

V. Determining the impact of such interventions, in a quantifiable manner, using validated instruments to assess perceptions of care coordination and self-efficacy, as well as monitoring concordance with guideline-recommended care by leveraging data from a network-wide decision support tool that captures systemic therapy selections.

OUTLINE:

Patients and caregivers receive access to the bladder cancer ENST and patients undergo psychological distress and nutrition screenings and may attend social work, psychology, and/or nutrition consultations as appropriate throughout the study. Patients, caregivers, and providers also attend virtual support group meetings periodically on study.

ELIGIBILITY:
Inclusion Criteria:

* PATIENTS: Age ≥ 18 years
* PATIENTS: Metastatic or locally advanced, unresectable bladder cancer
* PATIENTS: Receiving or planning to receive systemic therapy for bladder cancer at Roswell Park Comprehensive Cancer Center (RPCCC)
* PATIENTS: Subjects can be enrolled any time from initial diagnosis of advanced disease to within 8 weeks after initiation of first-line systemic therapy for advanced bladder cancer
* PATIENTS: Able to speak, understand, read, and write English
* CAREGIVERS: Age ≥ 18 years
* CAREGIVERS: Only caregivers of enrolled patients will be included in the study
* CAREGIVERS: Should be able to speak, understand, read, and write English
* CAREGIVERS: Caregivers will be enrolled in the study during the same time window as for patient enrollment (from initial visit to within 8 weeks of patients starting frontline therapy)

Exclusion Criteria:

* PATIENTS: Not receiving any form of systemic therapy for bladder cancer due to Eastern Cooperative Oncology Group (ECOG) performance status (PS) > 3, co-morbidities, or inadequate organ function
* PATIENTS: Predominantly small cell histology
* PATIENTS: Adults with impaired decision-making capacity, assessed by the study team to be unable to participate in ENST-based education and surveys
* PATIENTS: Pregnant women
* CAREGIVERS: Cognitively impaired adults/adults with impaired decision-making capacity
* CAREGIVERS: Individuals who are not yet adults (infants, children, teenagers)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-01-12 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Organizational readiness for implementing change (ORIC) | At baseline and at 6 months post-implementation
  A 12 item instrument used to determine how well employees feel they can implement the change in process .. Each item includes a scale from 1 (Disagree ) to 5 (Agree)
Guideline-concordant care at the institutional level | At baseline and at 6 months intervals for the study duration
  Guideline-concordant care at the institutional level will be calculated as the percentage of all systemic treatment decisions captured in the Clinical Oncology Pathway.
Patient perception of care coordination | At baseline and at 3 and 6 months post-implementation
  Patient perception of care coordination will be measured using Care Coordination Instrument.
Patient perception of self-efficacy | At baseline and at 3 and 6 months post-implementation
  Patient perception of self-efficacy will be measured using Generalized Self-Efficacy scale. A 10 item psychometric scale with 4 choice responses ranging from 1 (not at all true) to 4 (Exactly true).
Caregiver perception of care coordination | At baseline and at 3 and 6 months post-implementation
  Caregiver perception of care coordination will be measured using Care Coordination Instrument for Caregivers.

CONTACTS AND LOCATIONS:
Overall Officials: Saby George, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States